CLINICAL TRIAL: NCT03853746
Title: Evaluating the Effects of Short-term B-cell Depletion on Long-term Disease Activity and Immune Tolerance in Relapsing Multiple Sclerosis
Brief Title: Short-term B-cell Depletion in Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00201318
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ocrelizumab (Experimental): All participants will receive Ocrelizumab
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Patient will be treated with two courses of ocrelizumab (Ocrevus) for one year and then will stop the medication and will be monitored for the return of the disease activity. Those who experience return of the disease activity can go back on the medication.
  Other Names: Ocrevus

SUMMARY:
Several disease-modifying therapies (DMTs) have been shown to be effective in reducing the disease activity in patients with relapsing forms of multiple sclerosis (MS) but these treatments, often need to be used continuously for an unknown duration, rendering the long-term use extremely expensive. In addition, chronic administration of DMTs is often associated with undesirable side effects. Among these medications, B-cell depleting monoclonal antibodies might have the properties of an ideal group of medications: i) B-cell depleting antibodies have proven to be extremely potent in reducing or stopping the disease activity in relapsing MS, ii) B-cell depleting antibodies are very safe if used for a short period and use for a short duration may stop the inflammatory disease activity over long term, although current clinical practice and protocols are based on continuing B-cell depletion for an unknown period of time. Indeed, early phase clinical trials of rituximab and ocrelizumab suggested that a short course treatment with B-cell depleting antibodies can have long term effects and disease activity will not return even long after B-cell repopulation in the blood.

This long-term effect might be related to the specific pattern of B-cell tolerance defect in patients with MS and the potential of its normalization with B-cell depleting antibodies. By analyzing the reactivity of recombinant antibodies expressed from single B-cells, the investigators' collaborators have demonstrated that the pattern of B-cell tolerance defect is different in people with MS who only display an impaired removal of developing autoreactive B-cells in the periphery while central B-cell tolerance in the bone marrow is functional in most patients. In contrast, patients with rheumatoid arthritis (RA), type-1 diabetes (T1D) or Sjögren's syndrome (SS) show defective central and peripheral B-cell tolerance checkpoints. As a consequence, while anti-B-cell therapy does not correct defective early B-cell tolerance checkpoints in T1D and only temporarily slows down autoimmune processes before newly generated autoreactive B-cells likely induce patient relapse, the investigators postulate that the efficacy of B-cell depleting antibodies in MS may be linked to the B-cell depleting antibodies' normal central B-cell tolerance and the production of a normal B-cell and T-cell compartment after anti-B-cell therapy.

The investigators' goal is to provide proof-of-concept that a short duration of treatment with B-cell depleting antibodies can correct B-cell tolerance defects in MS and allow for medication-free prolonged freedom from disease activity, at least in a proportion of subjects with relapsing MS.

In an open label study, 10 patients with active relapsing MS will be treated with two courses of ocrelizumab and will be followed clinically and radiologically for at least two and a half years. Time to the return of disease activity (defined as clinical relapses or new or enhancing lesions on the MRI) will be the primary outcome of the study. The investigators will harvest B-cells before starting the treatment and after B-cell repopulation and assess the central and peripheral tolerance defects. The investigators hypothesize that in most participants, the disease activity will not come back, and this prolonged response to anti cluster of differentiation 20 (CD-20) therapy is associated with normalization of B-cell tolerance defect in these patients. Considering the safety of this approach, it can be adopted widely among people with MS. Hence, the proposed B-cell analyses before and after B-cell depletion in people with MS will provide novel insights regarding the mechanisms underlying the beneficial effect of B-cell depleting antibodies and the potential long-term suppression of disease activity. This strategy can therefore improve the approach to treatment of many people with relapsing MS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Diagnosis of relapsing-remitting multiple sclerosis (RRMS) based on revised McDonald criteria
* At least two Gd-enhancing lesions on the brain or spinal cord MRI done in the prior three months
* Naïve to disease modifying therapies or using an injectable therapy (interferons or glatiramer acetate); or, if history of receiving natalizumab, fingolimod, dimethyl fumarate and teriflunomide, no exposure for past three months
* Expanded Disability Status Scale (EDSS) score at the time of screening =<3

Exclusion Criteria:

* Contraindication to treatment with B-cell depleting antibodies, including being seropositive for HBsAg or HIV antibody or T-spot (or Quantiferon-Gold) positive
* Ever received B-cell depleting antibodies (rituximab, ocrelizumab, ofatumumab), alemtuzumab, daclizumab, mitoxantrone or hematopoietic stem-cell transplant
* Female who are pregnant, nursing or unwilling to use contraception up to six months after the second course of the infusion (or 12 months after the first infusion)
* Treatment with steroids in the past 30 days
* Clinically unstable medical or psychiatric disorders at the time of screening that require acute treatment as determined by the PI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, MD, MAS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Salazar-Camelo A, Vega L, Fadlallah Y, Bou Rjeily N, Balshi A, Morris B, Ghajarzadeh M, Mowry EM, Waubant E, Nourbakhsh B. Finite-course ocrelizumab in relapsing multiple sclerosis: Results of two prospective open-label trials with matched controls. Mult Scler. 2025 Oct;31(11):1338-1347. doi: 10.1177/13524585251375350. Epub 2025 Sep 19. PMID 40970353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ocrelizumab
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant dropped out immediately after signing the informed consent form and was not included in the subsequent analyses.
  years | 29.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Expanded Diability Status Scale [Median (Full Range); unit: points] — The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis, ranging from 0 (normal neurological exam) to 10 (death due to MS), with higher scores indicating greater disability.
  points | 2 [1 to 3]
Participants Who Received Prior Disease Modifying Therapy [Number; unit: Count]
  No medication | 7
  Glatiramer | 2
Disease Duration [Mean (Standard Deviation); unit: years] | 2.9 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Return of Disease Activity After the Third Month Post-first-infusion
Description: Number of patients with a return of disease activity after the third month post-first-infusion, objectively demonstrated by development of new T2 hyperintense lesions or Gd-enhancing lesions on the MRI or a clinical relapse that is confirmed with an objective change in the neurological examination.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 9
Participants
  Participants who experienced a return of disease activity | 3
  Participants who did not experience a return of disease activity | 6

2. Secondary Outcome: Change in Disability as Assessed by Expanded Disability Status Scale (EDSS)
Description: EDSS scores range from 0 to 10, with 0.5 steps. The higher the score, the worse the MS-related disability. Although the outcome was measured every six months, we used a linear mixed-effects model to analyze the data. The coefficient from this model represents the change in the outcome per unit of time (month), allowing for a consistent interpretation of the rate of change.
Time Frame: Every 6 months, up to 30 months
Measure: Mean (95% Confidence Interval); unit: Points change per month
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 9
Points change per month | -0.009 [-0.0183 to -0.0004]

3. Secondary Outcome: Change in a Quality of Life Measure as Assessed by Neuro-QoL Computer Adaptive Test (CAT) Fatigue Test
Description: The CAT produces a T-score (standardized score with a mean of 50 and a standard deviation (SD) of 10). A higher Neuro-QoL T-score represents more of the concept being measured. Here is the change in score from baseline to month 30. Although the outcome was measured every six months, we used a linear mixed-effects model to analyze the data. The coefficient from this model represents the change in the outcome per unit of time (month), allowing for a consistent interpretation of the rate of change.
Time Frame: Every 6 months, up to 30 months
Measure: Mean (95% Confidence Interval); unit: point chnage per month
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 9
point chnage per month | -0.012 [-0.15 to 0.12]

ADVERSE EVENTS:
Time Frame: Post last ocrelizumab treatment up to 24 months
Arm/Group | Ocrelizumab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=9)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT03853746/Prot_SAP_001.pdf